CLINICAL TRIAL: NCT05756478
Title: Appropriate Prescribing for Older Adults With Multimorbidity (Pro-M): A Feasibility Study
Brief Title: Appropriate Prescribing for Older Adults With Multimorbidity (Pro-M)
Acronym: Pro-M
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Geriatric Education and Research Institute (Other Government)
Collaborators: Tan Tock Seng Hospital (Other); Changi General Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: GERI1630
Record Dates: First submitted 2023-01-30; First posted 2023-03-06 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2024-02

CONDITIONS: Potentially Inappropriate Medications; Multimorbidity; Polypharmacy
Keywords: Inappropriate prescribing; Feasibility study
MeSH Terms: interventions — Medication Review

STUDY DESIGN:
Intervention Model Description: In order to investigate if implementing routine pharmacist-led medication reviews in the outpatient clinics of public hospitals for older adults with multi-morbidity, we are conducting a single-arm study at 2 sites to understand how the implementation strategies could be best carried out to facilitate the aim to reduce inappropriate prescribing. Pre- and post-medication review data on potentially inappropriate medications and other issues flagged will also be collected for a future scale up study. Each site is expected to recruit 30 patients.
  An evaluation will also be conducted with the doctors and pharmacists delivering and implementing the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Medication Review (Other): This is a feasibility study of implementing a pharmacist-led medication review using prescribing tools (e.g. STOPP/START, Beers Criteria) .
  Interventions: Other: Medication review

INTERVENTIONS:
Other: Medication review — This is a feasibility study of implementing a pharmacist-led medication review using prescribing tools (e.g. STOPP/START, Beers Criteria)

SUMMARY:
This is a two-site feasibility study to test implementation of an intervention that aims to reduce inappropriate prescribing for older adults with multimorbidity in geriatric medicine specialist clinics at public hospitals in Singapore. The specific aims are:

1. To assess the implementation outcomes: Appropriateness, Penetration/Reach, Acceptability, Feasibility, Sustainability (primary)
2. To collect data on recruitment and pre-post data on prevalence of potentially inappropriate prescribing (PIP) for the purpose of determining sample size for a scale up next phase study (secondary).
3. To conduct cost analysis of the intervention (secondary).

DETAILED DESCRIPTION:
The Appropriate prescribing for older adults with multi-morbidity (Pro-M) study aims to assess the feasibility of implementing routine medication review using prescribing criteria for older adults with multi-morbidity at the Geriatric Medicine outpatient clinics at 2 public hospitals in Singapore. The study will consist of a recruitment and implementation period and an evaluation period at the end.

Flow of the intervention (6 months):

1. Eligible patients with multimorbidity and are taking at least 5 medications daily will be identified and invited by the doctor to undergo medication review (MR).
2. Patients will undergo medication reviews with a pharmacist, involving the use of specific prescribing criteria and tools (e.g. STOPP/START, Beers Criteria), as determined by the sites.
3. Medication review findings will be documented in the electronic medical records and shared with the doctor, who will review the findings and make necessary changes to patients' prescriptions during consultations with the patients.
4. The Doctors will document the review outcome and prescribing decisions in the electronic medical records and communicate the changes (if any) to other relevant prescribers.
5. Patients will be invited to do a short survey on their experiences of the intervention at the end to assess implementation outcomes.

The intervention will be compared to 'usual care', where medication review is only done in an ad-hoc and informal basis. Patients' last consultation prior to the intervention period would be used as the point to measure 'usual care'.

Evaluation(3 months):

Doctors and pharmacists who implemented the study (delivery or support) will be invited to a survey and selected in-depth interviews to assess implementation outcomes.

ELIGIBILITY:
Inclusion Criteria for patients:

* Older adults age 65 and above
* Currently attending Geriatric Medicine Clinic
* on at least 5 medications.

Exclusion Criteria for patients:

* Those younger than 65
* Not a Geriatric Medicine outpatient clinic patient
* On fewer than 5 medications
* Currently receiving other pharmacist-related services such as medication therapy management.
* Non-English, non-Chinese, and non-Malay speaking patients.
* Patient or caregiver who declines any of the study procedure required within the intervention framework.

Inclusion Criteria for implementer:

* Doctors and pharmacists
* who are involved in the delivery or support of the intervention during the implementation period.

Exclusion criteria for implementer:

* Those who are not involved in the implementation of the study.
* Those who are not involved in the delivery of the intervention.

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-10-16 (Actual); Study Completion 2023-10-16 (Actual)

PRIMARY OUTCOMES:
Patients' attitudes towards acceptance of the intervention (Penetration/Reach) | A single-time-point survey to be administered immediately after the intervention
  The survey consists of 11 items, and each item is on a 5-point Likert scale (level of agreement). This is a mixed method implementation study that is focused on investigating the feasibility of implementing medication reviews as routine care for older adults with multimorbidity in the outpatient clinics. The first 6 months will be the implementation period, followed by a 3-month evaluation period that consists of a first survey of the implementers (doctors and pharmacists), then an in-depth interview with selected implementers.
Implementers' attitudes towards the appropriateness of the intervention | 3-month Evaluation period: A single-time-point survey to be conducted immediately after the 6-month implementation period. Selected in-depth interviews will follow to provide a qualitative context to the survey results.
  The survey consists of 25 items, and each item is measured on a 5-point Likert (level of agreement).
  This is a mixed method implementation study that is focused on investigating the feasibility of implementing medication reviews as routine care for older adults with multimorbidity in the outpatient clinics. The first 6 months will be the implementation period, followed by a 3-month evaluation period that consists of a survey of the implementers (doctors and pharmacists), then an in-depth interview with selected implementers.
Implementers' attitudes towards the acceptability of the intervention | 3-month Evaluation period: A single-time-point survey to be conducted immediately after the 6-month implementation period. Selected in-depth interviews will follow to provide a qualitative context to the survey results.
  The survey consists of 25 items, and each item is measured on a 5-point Likert (level of agreement).
  This is a mixed method implementation study that is focused on investigating the feasibility of implementing medication reviews as routine care for older adults with multimorbidity in the outpatient clinics. The first 6 months will be the implementation period, followed by a 3-month evaluation period that consists of a survey of the implementers (doctors and pharmacists), then an in-depth interview with selected implementers.
Implementers' attitudes towards the feasibility of the intervention. | 3-month Evaluation period: A single-time-point survey to be conducted immediately after the 6-month implementation period. Selected in-depth interviews will follow to provide a qualitative context to the survey results.
  The survey consists of 25 items, and each item is measured on a 5-point Likert (level of agreement).
  This is a mixed method implementation study that is focused on investigating the feasibility of implementing medication reviews as routine care for older adults with multimorbidity in the outpatient clinics. The first 6 months will be the implementation period, followed by a 3-month evaluation period that consists of a survey of the implementers (doctors and pharmacists), then an in-depth interview with selected implementers.
Implementers' attitudes towards the sustainability of the intervention. | 3-month Evaluation period: A single-time-point survey to be conducted immediately after the 6-month implementation period. Selected in-depth interviews will follow to provide a qualitative context to the survey results.
  The survey consists of 25 items, and each item is measured on a 5-point Likert (level of agreement).
  This is a mixed method implementation study that is focused on investigating the feasibility of implementing medication reviews as routine care for older adults with multimorbidity in the outpatient clinics. The first 6 months will be the implementation period, followed by a 3-month evaluation period that consists of a survey of the implementers (doctors and pharmacists), then an in-depth interview with selected implementers.
Implementers' views on the fidelity of the intervention. | :3-month Evaluation period: A single-time-point survey to be conducted immediately after the 6-month implementation period. Selected in-depth interviews will follow to provide a qualitative context to the survey results.
  The survey consists of 25 items, and each item is measured on a 5-point Likert (level of agreement).
  This is a mixed method implementation study that is focused on investigating the feasibility of implementing medication reviews as routine care for older adults with multimorbidity in the outpatient clinics. The first 6 months will be the implementation period, followed by a 3-month evaluation period that consists of a survey of the implementers (doctors and pharmacists), then an in-depth interview with selected implementers.

SECONDARY OUTCOMES:
Recruitment rate | 6 months during implementation period
  The rate will be measured by the number of participants enrolled in the intervention divided by the number of patients pre-screened as being eligible for the intervention. This information will inform sample size calculation for the next phase scale-up study.
  * Percentage of patients with at least one potentially inappropriate medication (PIM) before and after intervention
  * Percentage of patients with other medication issues identified before and after intervention.
Effectiveness of the intervention: Percentage of patients with at least one PIM before and after intervention. | 6 months during implementation period
  The rate will be measured by the number of patients prescribed with at least 1 PIM at the start of the intervention divided by total number of patients enrolled. It will then be compared to the rate of patients prescribed with at least 1 PIM after they had completed the intervention. This information will inform sample size calculation for the next phase scale-up study.
  • Cost of medications identified before and after medication review: cost of PIM and/or other medications issues identified will be collected during the implementation period.
Effectiveness of the intervention: Percentage of patients with other medication issues identified before and after intervention. | 6 months during implementation period
  The rate will be measured by the number of patients prescribed with at least 1 other medication issues at the start of the intervention divided by total number of patients enrolled. It will then be compared to the rate of patients prescribed with at least 1 other medication issues after they had completed the intervention. This information will inform sample size calculation for the next phase scale-up study.
Manpower cost to conduct medication review | 6 months during implementation period
  The cost would be measured by the estimated number of manpower hours needed to deliver the intervention multiplied by the manpower norm costs. This information will be utilized to calculate cost of implementing the intervention.
Cost of PIM and other medications with issues identified before and after medication review. | 6 months during implementation period
  The cost would be measured by calculating the subsidized cost of the identified medications (PIM and other medications with issues) prescribed to the enrolled patients. This information will be utilized to calculate cost of implementing the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Penny Lun, M.A., Principal Investigator — Geriatric Education and Research Institute, Singapore
Locations (2):
- Singapore (2):
  - Changi General Hospital, Singapore, Sinagpore
  - Tan Tock Seng Hospital, Singapore

REFERENCES:
- [Derived] Tang JY, Teng PHJ, Chen CY, Tan KT, Ang W, Lau S, Ang AGC, Kyaw KK, Tay XY, Lim WMS, Espeleta WDV, Lin H, Ding YY, Lun P. Appropriate Prescribing for older adults with Multimorbidity (Pro-M): protocol for a feasibility study. Arch Public Health. 2024 Mar 18;82(1):37. doi: 10.1186/s13690-024-01264-x. PMID 38500190